CLINICAL TRIAL: NCT04305561
Title: Comparison of CEUS With Conventional Ultrasound (US) to Dual-tracer 99mTcO4-/99mTc-MIBI Subtraction Scintigraphy With SPECT/CT for Localizing Pathological Parathyroid Glands in Patients With Primary Hyperparathyroidism
Brief Title: Preoperative Localization Strategies in Primary Hyperparathyroidism
Acronym: CEUS-project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Sanne Høxbroe Michaelsen, Principal Investigator, Odense University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: S-20190077
Record Dates: First submitted 2020-01-24; First posted 2020-03-12 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Primary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Intervention Model Description: Prospective paired cohort study.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound + Contrast-enhanced ultrasound (Other): Patients are offered a contrast-enhanced ultrasound (CEUS) examination in addition to conventional imaging. All included patients undergo both CEUS and conventional imaging, enabling them to act as their own controls.
  Pilot study: 60 patients Main study: 112 patients
  Interventions: Procedure: Contrast-enhanced ultrasound
- Conventional imaging (No Intervention): Dual-tracer 99mTechnetium-pertechnetate/ 99mTechnetium-sestamibi subtraction scintigraphy with single-photon emission computerised tomographic/CT fusion imaging (SPECT/CT) combined with conventional ultrasound.
  Pilot study: 60 patients Main study: 112 patients

INTERVENTIONS:
Procedure: Contrast-enhanced ultrasound — Ultrasound contrast agent: Stabilized sulfur hexafluoride microbubbles (SonoVue®, Bracco).
  An 18 G needle will be placed in an antecubital vein and directly attached to a three-way stopcock with an extension tube.
  The SonoVue® will be prepared and shaken shortly before injection in accordance with the instructions provided in the product information leaflet.
  The patient will be injected with 1.2 ml SonoVue® at a pace of 1-2 ml/s using the 180 degree straight-flow channel of the three-way stopcock, directly followed by a 10 ml bolus of sodium chloride 9 mg/mL (0.9%) injected into the 90 degree channel of the three-way stopcock at a pace of approximately 2 ml/s.
  A full examination will typically require one to two injections of 1.2 ml of SonoVue® (one injection per suspected parathyroid adenoma).
  Arms: Ultrasound + Contrast-enhanced ultrasound

SUMMARY:
The purpose of this project is to examine, in a non-inferiority study, whether the combination of conventional ultrasound and contrast-enhanced ultrasound (CEUS) can replace the radiation-based imaging modalities that are currently used to localize pathological parathyroid glands prior to surgical removal in patients with primary hyperparathyroidism.

This will take the form of a prospective paired cohort study where included patients receive a contrast-enhanced ultrasound examination in addition to the standard preoperative imaging regimen (subtraction scintigraphy with SPECT/CT and conventional ultrasound). Patients act as their own controls as all included patients undergo both CEUS and conventional imaging.

DETAILED DESCRIPTION:
The human body has four parathyroid glands. These are located in the neck at the backside of the thyroid gland. The four glands produce parathyroid hormone which regulates the amount of calcium in the blood. If one or more of the thyroid glands becomes hyperactive, too much parathyroid hormone is secreted into the blood. This condition is called hyperparathyroidism and results in elevated serum calcium levels. If left untreated, hyperparathyroidism may result in weak bones (osteoporosis), bone fractures, kidney stones and a myriad of unspecific symptoms.

In the vast majority of cases, only one of the four parathyroid glands is responsible for the disease, and the cure is surgical excision of the hyperactive gland. Such a surgery has traditionally involved a dissection of both sides of the neck, allowing the surgeon to visually inspect all four parathyroid glands to determine which gland(s) were hyperactive. Nowadays, if the hyperactive gland can be identified by parathyroid imaging prior to surgery, the surgeon can perform a minimally invasive procedure, focusing on the removal of a single gland. Such a focused procedure minimizes surgical risks and results in a shorter duration of surgery.

The parathyroid imaging regimen currently requires two out-patient visits on two separate days. The patient first visits the Department of Nuclear Medicine where a scan involving two radioactive tracers (a subtraction scintigraphy) and a 3D-examination (a SPECT/CT scan) are performed. The second visit takes place at the department of Head and Neck Surgery, where a head and neck surgeon performs an ultrasound examination of the neck.

The scans at the Department of Nuclear Medicine require the patient to lie completely still for a long time, expose the patient to some degree of radiation, and are relatively expensive. The ultrasound examination is fast and inexpensive, but isn't as sensitive as the scintigraphy (76% versus 70-92%).

Our project attempts to increase the sensitivity of the ultrasound examination by adding on an intravenous contrast agent. The contrast agent stays solely within the blood vessels, where it enhances the ultrasound signal. Contrast-enhanced ultrasound (CEUS) does not expose the patient to radiation, is fast to carry out, and the patient can be informed about the result of the scan immediately.

We hope that by introducing CEUS, we can change the order in which patients are examined prior to surgery, meaning that ultrasound - with or without an added contrast agent - will be the primary parathyroid imaging modality, and that patients will only continue to the Department of Nuclear Medicine if the result of the CEUS examination is uncertain.

Purpose

The purpose of this project is to examine, in a non-inferiority study, whether the combination of conventional ultrasound and contrast-enhanced ultrasound (CEUS) can replace the radiation-based imaging modalities that are currently used to localize pathological parathyroid glands prior to surgical removal in patients with primary hyperparathyroidism.

Method

This will take the form of a prospective paired cohort study where patients receive a contrast-enhanced ultrasound examination in addition to the standard preoperative imaging regimen (subtraction scintigraphy with SPECT/CT and conventional ultrasound). The CEUS examiner will be blinded to the results of the subtraction scintigraphy and SPECT/CT. The surgeon will have access to the results of all the preoperative imaging procedures, including CEUS. Correct localization of a hyperactive parathyroid gland on preoperative imaging is confirmed by a histological examination of the surgical specimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older with primary hyperparathyroidism (defined as an ionized calcium level above the upper reference level and a concomitant parathyroid hormone level in or above the upper third of the reference interval with no other known reason for the hyperparathyroid hypercalcemia) referred to the Department of ORL, Head and Neck Surgery at Odense University Hospital for parathyroidectomy.

Exclusion Criteria:

* Allergy to the contrast agent SonoVue®.
* Not legally competent.
* Does not read or speak Danish.
* Other causes of hypercalcemia (e.g. familial hypocalciuric hypercalcemia, pharmacologically or neoplastically induced hypercalcemia, secondary or tertiary hypercalcemia, uncontrolled hyperthyroidism, adrenal insufficiency, granulomatous diseases).
* Persistent or recurrent hyperparathyroidism.
* Previous surgery to the thyroid or the parathyroid glands.
* Current malignancy.
* Breastfeeding.
* Pregnancy.
* Contraindications to the use of SonoVue® (right-to-left shunts, severe pulmonary hypertension (pulmonary pressure >90 mmHg), uncontrolled systemic hypertension, adult respiratory distress syndrome, recent acute coronary syndrome, clinically unstable ischaemic cardiac disease within the last seven days, severe heart rhythm disorders, acute heart failure, or chronic heart failure class III or IV according to the New York Heart Association).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity of surgeon-performed conventional ultrasound | No residual disease 6 months after surgery
  With the histopathological result of the surgically removed specimen(s) as the reference standard, what is the sensitivity, specificity, positive and negative predictive value of the following imaging modalities in localising pathological parathyroid glands to the correct side, quadrant, and Odense Classification?
  a. Surgeon-performed conventional ultrasound
Sensitivity of contrast-enhanced ultrasound | No residual disease 6 months after surgery
  With the histopathological result of the surgically removed specimen(s) as the reference standard, what is the sensitivity, specificity, positive and negative predictive value of the following imaging modalities in localising pathological parathyroid glands to the correct side, quadrant, and Odense Classification?
  b. Surgeon-performed conventional ultrasound combined with contrast-enhanced ultrasound (CEUS).
Sensitivity of radiation based imaging | No residual disease 6 months after surgery
  With the histopathological result of the surgically removed specimen(s) as the reference standard, what is the sensitivity, specificity, positive and negative predictive value of the following imaging modalities in localising pathological parathyroid glands to the correct side, quadrant, and Odense Classification?
  c. Dual-tracer 99mTechnetium-pertechnetate/ 99mTechnetium-sestamibi subtraction scintigraphy (99mTcO4-/99mTc-MIBI) with single-photon emission computerised tomographic/CT fusion imaging (SPECT/CT).

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michaelsen SH, Bay M, Gerke O, Vestergaard S, Graumann O, Nielsen VE, Madsen AR, Bonnema SJ, Godballe C. Evaluation of Surgeon-Performed Ultrasonography With or Without Contrast Enhancement vs Scintigraphy in Patients With Primary Hyperparathyroidism. JAMA Otolaryngol Head Neck Surg. 2023 Jun 1;149(6):531-539. doi: 10.1001/jamaoto.2023.0389. PMID 37052913